CLINICAL TRIAL: NCT01663961
Title: An Open-label, One-sequence Crossover Study to Evaluate the Effect of Multiple Doses of YM178 on the Pharmacokinetics of Digoxin in Healthy Subjects
Brief Title: A Study to Evaluate the Effect of a Single Dose of Digoxin on the Actions in the Bodies of Healthy Subjects After Having Taken Several Doses of YM178
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 178-CL-059; 2008-000218-59 (EudraCT Number)
Record Dates: First submitted 2012-07-30; First posted 2012-08-14 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Healthy
Keywords: Phase I; Pharmacokinetics; YM178 Oral Controlled Absorption System (OCAS); Digoxin (Lanoxin); DDI (Drug-drug interaction); Open-label; Steady-state; subjects
MeSH Terms: interventions — mirabegron; Digoxin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- YM178 OCAS + digoxin (Experimental)
  Interventions: Drug: YM178 OCAS; Drug: Digoxin

INTERVENTIONS:
Drug: YM178 OCAS — oral
  Other Names: Mirabegron; Myrebtriq
Drug: Digoxin — oral
  Other Names: Lanoxin

SUMMARY:
A study that evaluates the interaction in healthy subjects of the heart drug Digoxin on YM178, when the latter is taken on a continuous basis, in order to establish that there is no risk to patients who may take this combination of drugs.

DETAILED DESCRIPTION:
Subjects receive a single oral dose of digoxin on Day 1. A full pharmacokinetic profile of digoxin is obtained for up to 144 hours post-dose. On the morning of Day 7, after the scheduled assessments are done, the subjects leave the clinic and return on Day 9.

From Day 10 up to and including Day 23, subjects receive daily oral doses of YM178 q.d. A single dose of digoxin is given in combination with YM178 on Day 18 (8 days after the first dose of YM178). On this day, a complete pharmacokinetic profile for digoxin is obtained up to 144 hours post-dose.

From Day 16 up to and including Day 19, blood samples for bioanalysis of YM178 are taken regularly. In addition, vital signs, safety ECG (Electrocardiogram) measurements, safety laboratory assessments, adverse events and concomitant medications are monitored throughout the investigational period.

Subjects return for a Post Study Visit 7-14 days after the last dosing occasion.

ELIGIBILITY:
Inclusion Criteria:

* Female subject must be of non-child bearing potential, i.e. post menopausal, surgically sterilized (e.g. tubal ligation), hysterectomy in medical history, or must practice an adequate (double barrier) non-hormonal contraceptive method to prevent pregnancies
* Body Mass Index ≥ 18.5 and < 30 kg/m2

Exclusion Criteria:

* History or presence of cardiac diseases, including arrhythmias (including 1st and 2nd degree atrioventricular heart blocks)
* History of hypokalemia, hypercalcemia or hypomagnesemia
* Any of the liver function tests (i.e. ALT, AST and Alkaline phosphatase) above the upper limit of normal at repeated measures
* Any clinically significant history of asthma, eczema, any other clinically significant allergic condition or previous severe hypersensitivity to any drug (excluding non-active hay fever)
* Any clinically significant history of gastrointestinal symptoms in the 4 weeks prior to admission to the clinical unit
* A marked baseline prolongation of QT/QTc interval after repeated measurements of > 450 ms, a history of unexplained syncope, cardiac arrest, unexplained cardiac arrhythmias or torsades de pointes, structural heart disease, or a family history of Long QT Syndrome (LQTS)
* Regular use of any inducer of liver metabolism (e.g. barbiturates, rifampin) in the 3 months prior to admission to the clinical unit
* Positive serology test for HBsAg, anti HAV (IgM), anti-HCV or anti-HIV 1+2

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2008-09; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To determine the effects of steady state YM178 levels on the pharmacokinetics (PK) of a single dose of digoxin | Pre-dose up to 144 hours post-dose
  Cmax (Maximum concentration), AUCinf (Area under the plasma concentration - time curve extrapolated until time = infinity)

SECONDARY OUTCOMES:
To evaluate the interaction between YM178 and digoxin in terms of safety and tolerability through assessment of adverse events, ECG and clinical laboratory assessments | Baseline to Post study visit (Up to 14 days after last dose)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Chair — Astellas Pharma Europe B.V.
Locations (1):
- SGS Aster, Paris, France